CLINICAL TRIAL: NCT05707780
Title: Clinical Evaluation of Resin Matrix Ceramic and Zirconia Posterior Crowns
Brief Title: Clinical Evaluation of Resin Matrix Ceramic Posterior Crowns
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Complutense de Madrid (Other)
Collaborators: BEGO GmbH (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UCM; 4195120 (Other Grant/Funding Number: BEGO GmbH)
Record Dates: First submitted 2023-01-22; First posted 2023-02-01 (Actual); Last update posted 2023-02-01 (Actual); Status verified 2023-01

CONDITIONS: Dental Materials
Keywords: crowns; monolithic zirconia; resin matrix ceramic; clinical evaluation; survival
MeSH Terms: interventions — Metal Ceramic Alloys

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Resin-matrix ceramic (Experimental): To assess the survival and clinical performance of resin-matrix posterior crows in a complete digital flow
  Interventions: Procedure: Resin-matrix
- Monolithic zirconia (Active Comparator): To assess the survival and clinical performance of monolithic zirconia posterior crows in a complete digital flow
  Interventions: Procedure: Monolithic zirconia
- Metal-ceramic (Active Comparator): To assess the survival and clinical performance of metal-ceramic posterior crows in a complete digital flow
  Interventions: Procedure: Metal-ceramic

INTERVENTIONS:
Procedure: Resin-matrix — posterior crowns
  Other Names: VarseoSmile crown
  Arms: Resin-matrix ceramic
Procedure: Monolithic zirconia — posterior crowns
  Arms: Monolithic zirconia
Procedure: Metal-ceramic — posterior crowns
  Arms: Metal-ceramic

SUMMARY:
The objectives of the present prospective randomized clinical study are to evaluate and to compare the survival and success rates, possible biological and technical complications, and the clinical performance of metal-ceramic, monolithic zirconia and resin-matrix posterior crowns.

The null hypothesis is that no differences would be found between the parameters studied for each type of restoration.

DETAILED DESCRIPTION:
A total of 60 patients, in whom the placement of a crown in the posterior region of the maxilla or mandible was indicated, will be included in the study. The patients will be recruited from the Master of Buccofacial Prostheses and Occlusion (School of Dentistry; University Complutense of Madrid). Prior to treatment, patients will be informed regarding the aims of the study, the clinical procedure, the materials used, the risks and benefits of ceramic restorations and the alternatives to the proposed treatment. All the patients will be provided with a written informed consent for the inclusion in this study, Ninety posterior crowns will be produced and assigned in parallel and randomly to either resin-matrix ceramic, zirconia or metal-ceramic restorations. Three experienced prosthodontists will treat the patients. Abutment preparation will be performed in a standardized manner: circumferentially chamfer (1 mm in width), axial reduction of 1 mm, and an occlusal reduction of 1.5 to 2 mm. The tapering angle between the axial walls will be approximately 10- to 12- degrees. Full-arch digital impressions will be taken using an Intraoral Scanner. The restorations will be cemented with a resin cement. The restorations will be examined at one week (baseline), 1, 2, and 3 years, by two researchers who were not involved in the restorative treatment

ELIGIBILITY:
Inclusion Criteria:

* One posterior tooth (molar or premolar) to be crowned,
* Vital abutments or abutments with sufficient endodontic treatment
* Abutment not crowned previously
* Periodontally healthy abutments with no signs of bone resorption or periapical disease --
* Adequate occlusogingival height
* Stable occlusion, and the presence of natural dentition in the antagonist arch.

Exclusion Criteria:

* Patients who present reduced crown length (less than 3 mm occlusogingival height
* Poor oral hygiene, high caries activity, active periodontal disease or bruxism.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-01-25 (Estimated); Primary Completion 2023-07 (Estimated); Study Completion 2026-10-30 (Estimated)

PRIMARY OUTCOMES:
Survival and success rates | 3 years
  Survival and success rates with Kaplan Meier method

SECONDARY OUTCOMES:
Quality of restorations at baseline | Baseline
  The restorations will be assessed using the California Dental Association's assessment system, for the surface and color, anatomic form, and margin integrity.
Quality of restorations at 1 year | 1 year
  The restorations will be assessed using the California Dental Association's assessment system, for the surface and color, anatomic form, and margin integrity.
Quality of restorations at 2 years | 2 years
  The restorations will be assessed using the California Dental Association's assessment system, for the surface and color, anatomic form, and margin integrity.
Quality of restorations at 3 years | 3 years
  The restorations will be assessed using the California Dental Association's assessment system, for the surface and color, anatomic form, and margin integrity.
Plaque Index (PI) at baseline | Baseline
  Plaque Index (PI) of the abutment and control tooth will be assessed. A score of 0 to 3 will be assigned. Higher score will mean a worse outcome
Plaque Index (PI) at 1 year | 1 year
  Plaque Index (PI) of the abutment and control tooth will be assessed. A score of 0 to 3 will be assigned. Higher score will mean a worse outcome
Plaque Index (PI) at 2 years | 2 years
  Plaque Index (PI) of the abutment and control tooth will be assessed. A score of 0 to 3 will be assigned. Higher score will mean a worse outcome
Plaque Index (PI) at 3 years | 3 years
  Plaque Index (PI) of the abutment and control tooth will be assessed. A score of 0 to 3 will be assigned. Higher score will mean a worse outcome
Gingival Index (GI) at baseline | Baseline
  Gingival Index (GI) of the abutment and control tooth will be assessed. A score of 0 to 3 will be assigned. Higher score will mean a worse outcome
Gingival Index (GI) at 1 year | 1 year
  Gingival Index (GI) of the abutment and control tooth will be assessed. A score of 0 to 3 will be assigned. Higher score will mean a worse outcome
Gingival Index (GI) at 2 years | 2 years
  Gingival Index (GI) of the abutment and control tooth will be assessed. A score of 0 to 3 will be assigned. Higher score will mean a worse outcome
Gingival Index (GI) at 3 years | 3 years
  Gingival Index (GI) of the abutment and control tooth will be assessed. A score of 0 to 3 will be assigned. Higher score will mean a worse outcome
Probing depth at baseline | Baseline
  Probing depth of the abutment and control tooth. A score of 0 to 4 will be assigned. Higher score will mean a worse outcome
Probing depth at 1 year | 1 year
  Probing depth of the abutment and control tooth. A score of 0 to 4 will be assigned. Higher score will mean a worse outcome
Probing depth at 2 years | 2 years
  Probing depth of the abutment and control tooth. A score of 0 to 4 will be assigned. Higher score will mean a worse outcome
Probing depth at 3 years | 3 years
  Probing depth of the abutment and control tooth. A score of 0 to 4 will be assigned. Higher score will mean a worse outcome
Margin stability at baseline | Baseline
  To assess the gingival margin stability of the abutment and control tooth throughout the evaluation period (subgingival, isogingival or supragingival)
Margin stability at 1 year | 1 year
  To assess the gingival margin stability of the abutment and control tooth throughout the evaluation period (subgingival, isogingival or supragingival)
Margin stability at 2 years | 2 years
  To assess the gingival margin stability of the abutment and control tooth throughout the evaluation period (subgingival, isogingival or supragingival)
Margin stability at 3 years | 3 years
  To assess the gingival margin stability of the abutment and control tooth throughout the evaluation period (subgingival, isogingival or supragingival)
Patient satisfaction at 3 years | 3 years
  Subjective patient satisfaction using Visual analogue scale (VAS) ranged from 0 (worst possile result) to 10 (best possible result)

CONTACTS AND LOCATIONS:
Overall Officials: MARIA JESUS SUAREZ, PhD, Principal Investigator — UNIVERSITY COMPLUTENSE OF MADRID; JESUS PELAEZ, PhD, Principal Investigator — UNIVERSITY COMPLUTENSE OF MADRID
Locations (1):
- Faculty of Odontology, Madrid, Spain